CLINICAL TRIAL: NCT05170152
Title: The Efficacy of Ultrasound Guided Corticosteroid Injection at A1 Pulley in Comparison to Percutaneous A1 Pulley Release as a Treatment for Idiopathic Trigger Finger
Brief Title: Ultrasound Guided Corticosteroid Injection at A1 Pulley in Comparison to Percutaneous A1 Pulley Release as a Treatment for Idiopathic Trigger Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: trigger finger
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: US-guided Release of the A1 Pulley Responsible for Trigger Finger is Feasible With a 21-gauge Needle

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- . Group A (Active Comparator): Underwent ultrasound guided methyl prednisolone acetate injection, between A1 pulley and tendons
  Interventions: Procedure: ultrasonography-guided injection
- Group B (Experimental): Underwent ultrasonography-guided percutaneous A1 pulley needle release
  Interventions: Procedure: pullae A1 release

INTERVENTIONS:
Procedure: ultrasonography-guided injection — ultrasonography-guided injection
  Arms: . Group A
Procedure: pullae A1 release — ultrasonography-guided pullae A1 release
  Arms: Group B

SUMMARY:
Objectives: To compare the efficacy of ultrasonography guided corticosteroid injection at A1 pulley and percutaneous A1 pulley release as a treatment for trigger finger.

Methods: 75 patients with idiopathic trigger finger were enrolled in our prospective study. Patients with diabetes mellitus, previous history of open release for trigger finger, different inflammatory arthritis and multiple trigger fingers affections were excluded. Group A 40 patients: Underwent ultrasound guided methyl prednisolone acetate injection, between A1 pulley and tendons .Group B 35 patients :Underwent ultrasonography-guided percutaneous A1 pulley needle release .All patients were subjected to the following before and after intervention by 1 and 3 months , DASH, trigger finger classification grade & VAS

DETAILED DESCRIPTION:
Trigger finger ( TF) is a pathologic problem of the finger leads to a painful tendon snap or click on flexion and extension, and/or locking of the metacarpophalangealor proximal interphalngeal joint (1) . Entrapment of the affected tendon at the first annular (A1) pulley occurs because of a differencein the diameter of the flexor tendon and its sheath as a result of thickening of the sheath and or localized tendon thickening.(1) . Most cases of trigger fingers are idiopathic and the incidence is around 28 cases per 100 000 population per year, or a lifetime risk of 2.6% in the general population and about 10% of patients are diabetics (1). Women are usually more affected than men, usually in the fifth and sixth decades(2) it is more common in women than in men, usually in the dominant hand, and most often in the thumb or ring fingers followed . (2) The diagnosis of trigger finger is based mainly on the medical history and clinical examination. The most important characteristic clinical sign is the mechanical blocking of the finger when flexed with painful snapping extended. (3). Management includes many options such as conservative treatment in the form of splinting, physical therapy, non-steroidal anti-inflammatory drugs, and local steroid injections, and surgical pulley release

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic trigger finger present for at least 3 months.

Exclusion Criteria:

* Patients with diabetes mellitus, previous history of open release for trigger finger, different inflammatory arthritis and multiple trigger fingers affections.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
trigger finger classification grade | 3 months
  trigger finger classification grade

SECONDARY OUTCOMES:
Pain score | 3 months
  visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
yes after publication